CLINICAL TRIAL: NCT06915324
Title: Transcranial Direct Current Stimulation (tDCS) of Brain Fog in Patients With Post Treatment Lyme Disease
Brief Title: Transcranial Direct Current Stimulation for Post Treatment Lyme Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Steven & Alexandra Cohen Foundation (Other)
Responsible Party: Principal Investigator, Brian A Fallon, Professor of Clinical Psychiatry, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAV1512; NCT06997341 (obsolete NCT alias)
Record Dates: First submitted 2025-04-02; First posted 2025-04-08 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Post-Treatment Lyme Disease
Keywords: tDCS; Cognitive training; Neuromodulation; Brain Fog; Brain Stimulation
MeSH Terms: conditions — Post-Lyme Disease Syndrome; Mental Fatigue | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Intervention Model Description: All participants receive computer-based cognitive exercises to improve processing speed. During the cognitive exercises, half of the participants receive concomitant active tDCS while the other half of the participants receive concomitant sham tDCS.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Cognitive training and active tDCS (Experimental): The cognitive training and brain stimulation sessions are conducted at home at the same time over 30 minutes, 5 days/week, for 4 weeks for a total of 20 sessions.
  Transcranial direct current stimulation (tDCS) is delivered by a user-friendly device; the participant wears a head-band that allows delivery of a weak electrical current (2mA) through two electrode patches over the forehead. The active stimulation session lasts 30 minutes.
  The cognitive training tasks are administered via a computer-based program BrainHQ (Posit Science). The BrainHQ adaptive cognitive training tasks have been previously associated with improved processing speed in other populations.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Cognitive training
- Cognitive training and sham tDCS (Sham Comparator): The cognitive training and brain stimulation sessions are conducted at home at the same time over 30 minutes, 5 days/week, for 4 weeks for a total of 20 sessions.
  Transcranial direct current stimulation (tDCS) is delivered by a user-friendly device; the participant wears a head-band that allows delivery of a weak electrical current (2mA) through two electrode patches over the forehead. The inactive (sham) stimulation session lasts 30 minutes.
  The cognitive training tasks are administered via a computer-based program BrainHQ (Posit Science). The BrainHQ adaptive cognitive training tasks have been previously associated with improved processing speed in other populations.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Cognitive training

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Transcranial direct current stimulation (tDCS) is delivered by a device that has a user-friendly interface and a large-button keypad, making it is easy to use at home. The device delivers a weak electrical current of 2.0 mA that is transmitted through two electrodes placed on the scalp to target the dorsolateral prefrontal cortex region of the brain. The electrodes are easily placed through a headset.
  The active stimulation session lasts 30 minutes.
  The inactive (sham) stimulation session will also last 30 minutes.
Behavioral: Cognitive training — The cognitive training tasks are administered via a computer-based program BrainHQ (Posit Science). There are 20 sessions, each 30 minutes a day, conducted over approximately 4 weeks. The BrainHQ adaptive cognitive training tasks have been previously associated with improved processing speed in other populations.

SUMMARY:
The primary purpose of this pilot study is to investigate a novel approach to the treatment of cognitive symptoms that persist despite prior antibiotic treatment for Lyme disease (Post treatment Lyme Disease or PTLD).

Aim 1: The primary aim of this study is to assess whether the processing speed of individuals with PTLD can be enhanced by combining transcranial direct current stimulation (tDCS) with computer based cognitive training games. To achieve this aim, over a 4-week period, all individuals with PTLD will participate in at home adaptive cognitive training combined with either active stimulation or sham stimulation.

Aim 2: To determine if treatment benefit in processing speed is sustained, the study will compare the sham and active groups 8 weeks after completion of study treatment.

DETAILED DESCRIPTION:
The primary purpose of this pilot study is to investigate a novel approach to the treatment of cognitive symptoms that persist despite prior antibiotic treatment for Lyme disease (Post treatment Lyme Disease or PTLD).

Processing speed has been shown to be one of the primary areas of cognition affected by PTLD and may be a critical component of "brain fog," an everyday term for the fuzzy/scattered thinking, lack of mental sharpness and forgetfulness commonly reported by PTLD patients. Deficits in processing speed may also relate to fatigue and have broader effects on other aspects of cognitive performance including problems with memory and language.

This study will enroll participants with PTLD (definitive, probable, possible) who will be randomly assigned to one of two treatment groups at a 1:1 ratio. The at-home treatment duration is 30 minutes daily for 20 sessions spanning approximately 4 weeks. Group 1 will receive active transcranial direct current stimulation (tDCS) combined with computer-based cognitive training. Group 2 will receive sham tDCS combined with computer-based cognitive training. The cognitive training exercises are personalized to each user's performance level and are aimed at improving cognitive performance by improving information processing speed.

The study will assess changes in cognitive functioning in the context of tDCS treatment using both formal neuropsychological tests as well as questionnaires regarding cognitive lapses in everyday situations. In addition, the study will be examining whether tDCS will lead to improvements in other aspects of functioning such as mood, fatigue and pain symptoms as measured by clinical rating scales.

ELIGIBILITY:
Inclusion Criteria:

* History of diagnosis of Lyme disease by a health care provider, meeting criteria for either definite or probable or possible LD
* Willingness to provide documentation of prior LD testing and/or related medical records
* Total prior antibiotic treatment for LD was at least 2 courses of antibiotic therapy
* Have cognitive symptoms attributed to Lyme disease that have persisted or returned despite antibiotic therapy
* Current cognitive symptoms interfere with function and/or cause distress
* Have evidence of slowed processing speed on a screening measure
* Participant is willing to be off of antibiotic treatment for tick-borne disease for at least 4 weeks prior to final determination of study eligibility and for the duration of the 12-week study.
* Participant expresses willingness to not start new medications that might affect treatment outcome during the trial (unless medically necessary), and willingness to inform study staff regarding any changes in medication
* Live in the US or Canada and comfortable speaking English
* Age 18-65
* Stable and continuous access to internet service
* Adequate home facilities (enough space, access to quiet and distraction free area)
* Able to commit to the 12-week study period (4 weeks of training sessions and an 8-week post treatment visit)
* Estimated intellectual ability >= 85

Exclusion Criteria:

- Medical Illness: Any of the following: a. Unstable non-Lyme-related chronic medical illness over the last 12 months (e.g., cancer, acute myocardial infarction, labile hypertension) b. Any severe skin disorder or skin sensitive area near stimulation locations (e.g. forehead)

Neurologic: Any of the following:

* History of traumatic brain injury with persistent post-concussive symptoms
* History of seizure disorder or recent (<5 years) seizure history
* History of neurosurgery to the head
* Chronic headaches or migraines of moderate to severe intensity within the last month
* Post stroke deficits that may interfere with assessment
* Any progressive neurodegenerative disorder or other neurological disorders that may interfere with assessment at discretion of the investigator.

Psychiatric: Any of the following:

* History of intellectual disability, or other developmental neurological condition associated with cognitive impairment
* Current primary psychiatric disorder that would interfere with ability to participate
* Current alcohol or other substance use disorder
* Current suicide risk as assessed by the C-SSRS (any level)
* History of suicidal behavior over the last year
* History of a diagnosis of a psychotic disorder, mania or bipolar disorder
* Depression rating of moderate or severe at screening

  * Currently taking opiate-based medications, dissociative drugs (prescribed or illicit), or other medication considered likely to interfere with treatment outcome at the discretion of the investigator. The use of a stable dose of benzodiazepines, anticholinergic agents and non-narcotic pain medications is permitted. The use of an occasional dose of these medications is also permitted, but not within 48 hours of neurocognitive study assessments.
  * Participants whose current daily medication regimen has not been stable for a minimum of 4 weeks prior to final determination of study eligibility
  * Medical device implanted in the head (such as a Deep Brain Stimulator) or in the neck (such as a Vagus Nerve Stimulator), or metal implants in the head or neck
  * Inadequate visual or motor skills needed for regular computer use or to operate study equipment, or inability to provide informed consent
  * Individuals who are pregnant or breastfeeding or planning to become pregnant
  * Lifestyle Considerations: Participants not willing to refrain from beginning, resuming or increasing non study cognitive training or cognitive enhancing supplements/medications or other therapies that might affect treatment outcome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Coding test scale score for acute treatment | 4 weeks
  The WAIS-IV Coding test is part of the Processing Speed Subtest and consists of three measured abilities, including visual-motor coordination, motor and mental speed, and visual working memory. In this coding task, participants using the key provided at the top of the exercise form draw the symbol under the corresponding number. Subtests yielding scaled scores that sum to derive the full-scale score. The score is the number of correct symbols from 0-133 drawn within a period of 120 seconds. The standardized T-score ranges from 1 to 19 with higher numbers indicating a better outcome/performance.
Coding test scale score for post-treatment follow-up | 12 weeks
  The WAIS-IV Coding test is part of the Processing Speed Subtest and consists of three measured abilities, including visual-motor coordination, motor and mental speed, and visual working memory. In this coding task, participants using the key provided at the top of the exercise form draw the symbol under the corresponding number. Subtests yielding scaled scores that sum to derive the full-scale score. The score is the number of correct symbols from 0-133 drawn within a period of 120 seconds. The standardized T-score ranges from 1 to 19 with higher numbers indicating a better outcome/performance.

SECONDARY OUTCOMES:
Composite score of the reaction time measures | 4 weeks
  Composite score of the reaction time measures (Coding, Choice Reaction Time, Grooved Pegboard, and the Test of Silent Word Reading Fluency-2), measured in Z-scores from -4 to +4 with a higher score representing a better outcome.
Fatigue Severity Scale (FSS) Score | 4 weeks
  This is a self-reported measure of fatigue. This measure consists of 9 items inquiring about the severity of fatigue in different situations over the past week. Scores for each item range from 1 to 7 where 1 indicates strong disagreement and 7 strong agreements. Higher scores indicate higher levels of fatigue.
General Symptom Questionnaire (GSQ-30) Score | 4 weeks
  This is a 30 item self-reported measure of symptom burden. The measure asks participants to rate how bothered they have been with a particular symptom over a 2-week time frame. The total score ranges from 0 to 120 with higher score indicating higher symptom severity.
Generalized Anxiety Disorder-7 (GAD-7) Score | 4 weeks
  This is a measure of severity of anxiety. It has 7 seven items, and the scores range from 0 to 21 with higher scores indicating more pronounced anxiety.
PROMIS Emotional Distress-Depression-Short Form Score | 4 weeks
  This is a self-reported measure that assesses symptoms of depression during the past 7 days. It has 8 items. Each item ranges from 1 (never) to 5 (always) with higher scores representing more pronounced depression.
Patient-Reported Outcomes Measurement Information System (PROMIS-29) symptom summary score | 4 weeks
  The PROMIS-29 is a 29 item self-report measure covering 7 symptom domains. The questions are ranked on a 5-point Likert Scale. The PROMIS-29 SPADE score represents the average T-score across the 5 SPADE (sleep disturbance, pain, anxiety, depression, and low energy/fatigue) domains with higher scores indicating greater symptom severity. The SPADE T-score ranges from 20-80 with higher scores indicating more symptom severity.
Cognitive functioning z-score | 4 weeks
  Measures that include domains of cognitive function that are affected by processing speed (attention, memory, working memory and language fluency). Each measure has a raw score that is converted to z-score that ranges from -4 to +4 with higher score representing a better outcome.
Neuro-QoL Short Form v1.0 - Applied Cognition Score | 4 weeks
  This is a self-reported measure that assesses cognitive function across neurological conditions. Items are scored on a 5-point scale that uses different language depending on assessment. The questions range from least (1) to most (5) based on frequency of behavior, amount of difficulty, or degree of agreement. Raw scores are converted based on consistent metric (T-distribution) with data from the US general population with a T-score mean of 50 and standard deviation of 10. Higher score indicates a greater degree of reported cognitive difficulties.
Brain Fog Visual Analogue Scale (Brain Fog VAS) Score | 4 weeks
  This is self-reported measure of cognitive complaints severity (brain fog). It measures the period over the last 7 days, score ranges from 0 to 10 with higher score indicating a higher severity of reported brain fog.

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Fallon, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Columbia University Department of Psychiatry, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided